CLINICAL TRIAL: NCT03697759
Title: A Decision Support System for Self-management of Low Back Pain - PILOTSTUDY
Acronym: selfBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Norwegian University of Science and Technology (Other); National Research Centre for the Working Environment, Denmark (Other Government); University of Glasgow (Other); Robert Gordon University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20182000-24; 2018/791 (Other: The Regional Committee for Medicine and Health Related Research Ethics)
Record Dates: First submitted 2018-08-10; First posted 2018-10-05 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
Keywords: Digital Decision Support System; App; Self-management
MeSH Terms: conditions — Low Back Pain; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This study is a pilot study preceding a randomized controlled trial. In the pilot study all enrolled participants are offered the intervention.
Masking Description: Since there is no randomization, all participants receive the intervention. Consequently, there is no blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual care + selfBACK (Experimental): Participants will use the selfBACK system and app
  Interventions: Other: Usual care + selfBACK

INTERVENTIONS:
Other: Usual care + selfBACK — The selfBACK intervention is a digital Decision Support System (DSS) for self-management of LBP provided to the participant via a smartphone app (selfBACK app). In addition, the participant is provided with a step-detecting wristband (Xiaomi Mi Band 2) that interacts with the selfBACK app.
  The DSS provides individually tailored self-management plans including content from three categories; 1) information/education, 2) physical activity monitoring through wearing the step-detecting wristband, and 3) strength and flexibility exercises. The weekly plans are individually tailored to the specific patient, using the data available from the patient, and each week the patients report back their progress on physical activity (step count) and exercise (volume completed). These data are matched with the patients follow-up data to create a self-management plan that is up to date and adaptable to variation in health-status of the individual patient.
  Other Names: selfBACK digital decision support system

SUMMARY:
The pilot study precedes a larger randomized controlled trial, to be starting in February 2019.

In this pilot study all participants are allocated to the intervention group.

The intervention consists of a digital decision support system delivering a weekly plan of suggested activities that the participant can use to self-manage their low back pain. The plan is presented to the participant in the selfBACK app.

DETAILED DESCRIPTION:
The selfBACK intervention consists of the selfBACK system, that provides the participants with an individually tailored weekly plan of suggested activities to use in their self-management of low back pain.

The SELFBACK system constitutes a data-driven predictive decision support system that uses Case-Based Reasoning methodology to capture and reuse participant cases in order to suggest the most suitable self-management plan for participants. The selfBACK system is an intelligent system that will adjust the suggested self-management plan to the individual participants by using the information available on the participant (baseline questionnaires), weekly self-reported of changes in health status through the app, and data on physical activity via the step-detecting wristband.

The weekly plan includes three categories of content; 1) information/education, 2) physical activity monitoring through wearing a step-detecting wristband, and 3) strength and flexibility exercises.

ELIGIBILITY:
Inclusion Criteria:

* Seeking care from primary health-care practice or a specialised outpatient hospital facility (DK) for non-specific LBP within the past 8 weeks
* LBP of any duration
* Mild-to severe pain-related disability rated as 16 or below on the PROMIS-PF4 function scale.
* Age: ≥18 years
* Own and regularly use a smart phone (with at least Android 7.0 or iOS11.0) with internet access (Wi-Fi and/or mobile data)
* Have a working email address and have access to a computer with internet access to complete questionnaires in a web browser.

Exclusion Criteria:

* Not interested
* Unable to speak, read or write in the national language (Danish/ Norwegian)
* Cognitive impairment or learning disabilities
* Pathology, such as fracture, cancer, inflammatory diseases, and signs of radiculopathy (severe leg pain, loss of leg strength, or loss of or altered sensation in a myotomal or dermatomal distribution)
* Serious mental illness, such as major depression, schizophrenia, and psychosis
* Terminal illness
* Unable to take part in exercise/physical activity (such as non-ambulatory patients, use of walking aids/assistance, unable to get down and up from the floor independently)
* Fibromyalgia (diagnosed by a Health Care Professional)
* Pregnancy
* Previous back surgery
* Ongoing participation in other research trials for LBP management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | change from baseline to 6 weeks
  The primary outcome is the Roland Morris Disability Questionnaire (RMDQ) assessing pain-related disability. The questionnaire includes 24 items asking participants to indicate if they experience functional impairments by answering "yes" or "no" to a series of descriptions of functional abilities with higher scores indicating higher level of disability.

SECONDARY OUTCOMES:
Pain intensity | change from baseline to 6 weeks
  Pain intensity measured as average and worst within the past week. Measured on a 0 - 10 Numerical Rating Scale with 0 being no pain and 10 being worst pain imaginable.
  Pain duration measures patients' selfreported length of current pain episode. Pain medication measures the frequency of the non-prescription pain medication use for low back pain.
The Fear avoidance Belief Questionnaire | change from baseline to 6 weeks
  The FABQ is a 5-item questionnaire, where the participants score their beliefs about their LBP on an ordinal scale ranging from zero [completely disagree] to six [completely agree]
Pain Self-Efficacy Questionnaire | change from baseline to 6 weeks
  The questionnaire assesses the participant's level of confidence in carrying out specific activities despite their pain [52, 53]. The PSEQ is a 10-item questionnaire scored on an ordinal scale ranging from zero [completely disagree] to six [completely agree].
Activity limitation | change from baseline to 6 weeks
  Activity Limitation evaluates if LBP has limited work and leisure time activities. The questionnaire consists of two single items with response options "yes" and "no".
Workability | change from baseline to 6 weeks
  Work Ability is measured by a single-item and rated on an 11-point NRS scale ranging from zero [completely unable to work] to 10 [work ability at its best].
Saltin-Grimby Physical Activity Level Scale | change from baseline to 6 weeks
  Participants indicate their amount of time per week performing leisure activities with four levels of intensity ranging from sedentary to vigorous physically active
Patient Specific Functional Scale | change from baseline to 6 weeks
  Participants rate their function on up to two self-selected activities, are asked to rate if they are unable to do or are having difficulty with the their ability to perform self-selected activities regarded as important by the participants themselves
Sleep | change from baseline to 6 weeks
  Sleep is assessed by self-report using four items concerning problems with falling asleep, waking up repeatedly, waking up too early, and feeling sleepy during the day.
Perceived Stress Scale | change from baseline to 6 weeks
  a 10-item questionnaire asking about frequency of thoughts and feelings related to perceived stress
Health-related Quality of Life | change from baseline to 6 weeks
  The EuroQoL 5-dimension (EQ-5D) questionnaire is used to asses quality of life within each of the five dimension (i.e., mobility, self-care, activities, pain/discomfort and anxiety/depression).
Brief Illness Perception Questionnaire | change from baseline to 6 weeks
  the questionnaire evaluates the participants' illness perception in an 8-item questionnaire. Items are scored on an ordinal scale ranging from zero [no problems] to 10 [worst severity].
Patient Health Questionnaire-8 | change from baseline to 6 weeks
  the questionnaire is an 8-item questionnaire used to evaluate the participants' depressive symptoms. Items are scored on a 4-point Likert scale scoring frequency of experiencing symptoms of depression.
Patients Global Perceived effect | 6 weeks
  a single item question for Patient's Global Perceived Effect will be asked at follow-up, where participants are asked to rate improvement or deterioration of their LBP compared to before the intervention
Patient Acceptable Symptom State | 6 weeks.
  a single item question on whether or not the patient considers their current symptom state as acceptable or not
Virtual Care Climate Questionnaire | 6 weeks
  The Virtual Care Climate Questionnaire concerns patients' perceived support for autonomy in a virtual care setting.
User ratings | 6 weeks
  Three rating questions on overall rating, ease of use and recommendation to others scored on a 5-point system

OTHER OUTCOMES:
Tailoring variables | Weekly for 6 weeks
  Participants in the intervention are on a weekly basis asked a set of tailoring questions. These are tracked over the intervention period. The tailoring questions include items on pain (NRS for pain intensity), function, fear-avoidance, work ability, sleep, pain self-efficacy, stress, symptoms of depression, and barriers for self-management.
  Note. not all questions are asked on a weekly basis
Physical activity | weekly for 6 weeks
  The patients' weekly recommended step count goal, and the actual achieved step count per. day
Exercise volume | weekly for 6 weeks
  The patients report back their completed exercise volume as number of set and repetitions for their suggested exercises, when they perform them

CONTACTS AND LOCATIONS:
Overall Officials: Karen Søgaard, PhD, Principal Investigator — University of Southern Denmark
Locations (2):
- Physical Activity and Health at Work, Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark
- Norwegian University of Science and Techonology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bach K, Szczepanski T, Aamodt A, Gundersen OE, Mork. PJ. Case Representation and Similarity Assessment in the selfBACK Decision Support System ICCBR 2016: Case-Based Reasoning Research and Development pp 32-46
- [Derived] Sandal LF, Overas CK, Nordstoga AL, Wood K, Bach K, Hartvigsen J, Sogaard K, Mork PJ. A digital decision support system (selfBACK) for improved self-management of low back pain: a pilot study with 6-week follow-up. Pilot Feasibility Stud. 2020 May 23;6:72. doi: 10.1186/s40814-020-00604-2. eCollection 2020. PMID 32489674
- See also: project webpage — http://www.selfback.eu